CLINICAL TRIAL: NCT02931903
Title: The Effect of Lithium Disilicate Glass-ceramic (IPS Emax) Versus Hybrid Ceramic (Vita Enamic) Superstructure Materials on Implant Stability in Implant Supported Restorations
Brief Title: Lithium Disilicate Glass-ceramic Versus Hybrid Ceramic Superstructure Materials on Implant Stability
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sally Edward Fekry, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: CEBD-CU-2016-10-219
Record Dates: First submitted 2016-10-11; First posted 2016-10-13 (Estimated); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Prosthesis Survival
Keywords: implant supported restorations; IPS Emax (lithium disilicate glass-ceramic); Vita Enamic (hybrid dental ceramic); implant survival; peri-implant tissue response
MeSH Terms: conditions — Prosthesis Failure | interventions — VITA Enamic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hybrid superstructure (Experimental): Vita Enamic is a hybrid ceramic, consisting of composite and ceramic. The ceramic; compatible and high aesthetics while the composite; resilient material with low modulus of elasticity which will absorb stress and therefore decrease load on bone and eventually decrease crestal bone loss
  Interventions: Other: Vita Enamic (hybrid dental ceramic)
- Ceramic superstructure (Active Comparator): IPS Emax, is the mostly used ceramic superstructures in implant supported restorations.
  Interventions: Other: lithium disilicate glass-ceramic

INTERVENTIONS:
Other: Vita Enamic (hybrid dental ceramic) — Vita Enamic (hybrid dental ceramic) are provided as blocks to be milled using Computer aided design/Computer aided manufacturer (CAD/CAM) technology,
  Other Names: hybrid, resin nanoceramic
  Arms: Hybrid superstructure
Other: lithium disilicate glass-ceramic — All ceramic crowns (Lithium disilicate glass ceramic) milled by Computer aided design/Computer aided manufacturer (CAD/CAM) technology
  Other Names: Emax CAD, IPS Emax
  Arms: Ceramic superstructure

SUMMARY:
The aim of this study is to assess the effect of the newly introduced (hybrid dental ceramic) superstructure materials, Vita Enamic versus IPS Emax on implant stability, patient satisfaction and crestal bone loss.

DETAILED DESCRIPTION:
This study will be conducted on patients requiring single implant replacement in the maxillary premolar area, admitted to the Outpatient Clinic of Fixed Prosthodontics Department, Faculty of Oral and Dental medicine, Cairo University.

After a period of healing of 6 months, an implant abutment of accurate diameter and angulation will be placed to fit precisely into the internal hex of the fixture after removal of the cover screw. The platform matched abutment will be then secured into its final position using the abutment screw. Alginate impression will be taken and poured into dental stone. Using the impression transfers, impressions with polyvinylsiloxane are taken. After taking the impressions, the Impression transfers are removed and fixed to the implant replica.

Surgeons' assistants will be asked to open the sealed envelope containing the information regarding the crown placement. The impressions will be sent to dental laboratory with the result of the sealed envelope, for preparation of the future crowns, either vita enamic crowns or Ips e max crowns.

ELIGIBILITY:
Inclusion Criteria:

Patients > 18 yrs. Patients with missing teeth in the maxillary premolar region. Absence of any pathological condition in the recipient site.

Stabilization phase will be performed including:

* Scaling
* Debridement.
* Elimination of all carious cavities and root canal treatment if needed.
* Elimination of over-hanging restoration. Systemic condition of the subjects was evaluated according to dental modification of the Cornell medical index (Kerr and Millard 1966).

Patients who are cooperative, motivated, and hygiene conscious. Patients should have adequate ridge width (>5mm).

Exclusion Criteria:

Patients unable to undergo minor surgical procedure. Patients with history of drug abuse or metabolic drugs. Patients with history of psychiatric disorder. Patients with insufficient bone. Patients with insufficient vertical inter-arch space, upon centric occlusion, to accommodate the available restorative components.

Patients with any systemic condition that may contraindicate implant therapy. Patients that may have any habits that may jeopardize the osseo-integration process, such as heavy smoking and alcoholism.

Patients with para-functional habits that produce overload on the implant such as bruxism and clenching.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01; Primary Completion 2017-12 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Implant survival rate | 12 months
  Implant stability and success could be affected by crestal bone loss, if the implant is stable therefore high survival rate

SECONDARY OUTCOMES:
Crestal bone loss | 12 months
  Crestal bone loss will be measured using a Cone Beam Computed tomography to measure the amount of bone resorbed from start date, and follow up for one year
Peri-implant tissue response | 12 months
  Bleeding index, probing depth and gingival index
Patient satisfaction | 12 months
  Patients will be asked to answer a questionnaire to know whether the procedure was not satisfied, accepted, or highly satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Gihan El Naggar, Professor, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: No